CLINICAL TRIAL: NCT02147730
Title: ALICE-Regional Anesthesia in Italy: Complications and Outcomes
Acronym: ALICE
Status: Completed | Type: Observational
Sponsor: Fondazione IRCCS Policlinico San Matteo di Pavia (Other)
Responsible Party: Principal Investigator, Massimo Allegri, MD, Fondazione IRCCS Policlinico San Matteo di Pavia
Other Study IDs: PT-SM-12-Alice
Record Dates: First submitted 2014-04-01; First posted 2014-05-28 (Estimated); Last update posted 2017-03-03 (Actual); Status verified 2017-03

CONDITIONS: Chronic Pain
Keywords: chronic pain
MeSH Terms: conditions — Chronic Pain | interventions — Anesthesia, Conduction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- surgical patients: all surgical patients undergoing gastrectomy, knee-hip-shoulder arthroplasty, hallux valgus surgery, hernia repair, saphenectomy, cesarean section,colectomy, hysterectomy, nephrectomy mastectomy during study period
  Interventions: Procedure: regional anesthesia; Procedure: non-regional anesthesia

INTERVENTIONS:
Procedure: regional anesthesia — all patients receiving a regional anesthesia/analgesia technique
Procedure: non-regional anesthesia — all patients receiving other-than-regional anesthesia techniques

SUMMARY:
Regional anesthesia techniques, with administration of local anesthetics for neuraxial or peripheral route are now playing a central role in modern anesthesia and in particular in the control of postoperative pain. There are many review and meta-analyzes suggesting that a good pain control, and specifically loco regional analgesia, may improve the outcome of patients undergoing surgery.

The control of acute post-operative pain is not the only challenge to be paid by anesthesiologists, because there is still much to be understood in relation to persistent post-surgical pain (PPP), and about the degree of influence that regional anesthesia plays in complete long-term functional recovery of patients.

From the pathophysiological perspective there is not a precise definition of the mechanisms and risk factors that determine the onset of the persistent pain after surgery, but, more in general, it seems to be related to a malfunction of the mechanism of secondary hyperalgesia.

Regional anesthesia could play a key role, as the main determinant of chronic pain is acute post-operative pain. The techniques of regional anesthesia exert a powerful block at the peripheral level, potentially preventing the progression of central pain and the persistence of stimuli that can reach the central nervous system. In addition, during surgery, these techniques can reduce the metabolic alterations and the triggering mechanisms of local and systemic pro-inflammatory mediators' release.

Few perspective studies exist about the influence of regional anesthesia on long-term outcome and persistent pain after surgery.

The objective of the investigators study is to assess in a prospective fashion the role of regional anesthesia/analgesia technique in preventing (or not) persistence pain occurrence after surgical interventions which are mostly associated to pain persistence, and understand if regional anesthesia provides advantages in other post-surgical outcomes.

ELIGIBILITY:
Inclusion Criteria:

* more than 18 ys old
* informed consent

Exclusion Criteria:

* reintervention
* ASA (American Society of Anesthesiologists) status 4 and 5
* emergency surgery
* no informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: all surgical patients undergoing gastrectomy, knee-hip-shoulder arthroplasty, allux valgus surgery, hernia repair, safenectomy, cesarean section,colectomy, hysterectomy, nephrectomy mastectomy during study period
Sampling Method: Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2013-01 (Actual); Primary Completion 2016-05 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Persistent Pain | 6 months
  prevalence of pain at 6 months after surgery. Pain will be assessed with NRS (Numeric Rating Scale) from 0 (no pain) to 10 (worst pain possible).

SECONDARY OUTCOMES:
Patients satisfaction | 6 months
  Patient satisfaction will be assessed with a verbal rating scale from 0 (completely dissatisfied) to 10 (completely satisfied).
quality of life | 6 months
  changes in quality of life after surgery will be assessed with a 5-point scale (very inferior, inferior, same of preoperatively, superior, very superior)
side effects | 6 months
  infection (local or systemic), postoperative neurologic symptoms, thrombotic events, post-dural puncture headache, postoperative nausea and vomiting, perforation/leakage, respiratory failure, heart failure, reintervention, death.
functional activity | 6 month
  expressed as number of days after the intervention before the patient has returned to a normal activity

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesia and ICU - IRCCS Policlinico S Matteo, Pavia, Pavia, Italy

REFERENCES:
- [Derived] Bugada D, Allegri M, Gemma M, Ambrosoli AL, Gazzerro G, Chiumiento F, Dongu D, Nobili F, Fanelli A, Ferrua P, Berruto M, Cappelleri G. Effects of anaesthesia and analgesia on long-term outcome after total knee replacement: A prospective, observational, multicentre study. Eur J Anaesthesiol. 2017 Oct;34(10):665-672. doi: 10.1097/EJA.0000000000000656. PMID 28767456